CLINICAL TRIAL: NCT03744052
Title: Using Neuroscience to Optimize Digital Health Interventions Across Adulthood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Duke University: Bass Connections (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00100499
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Participants (Experimental): Messages regarding physical activity will be texted to participants.
  Interventions: Other: Motivational Messages

INTERVENTIONS:
Other: Motivational Messages — Messages regarding physical activity will be texted to participants.

SUMMARY:
The goal of this study is to investigate the extent to which brain imaging data predict health behavior change, compared to participant self-reports.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 30-80 who read/understand English, 50% male and 50% female, and a maximum of 50% will be white.

Exclusion Criteria:

* Pregnancy
* History of head injury
* Mental illness diagnosis
* Psychoactive medication
* Psychiatric or neurological history
* Claustrophobia
* Ferrous metal implanted within the body (those with fMRI-compatible implanted devices will not be excluded, but the eligibility of their devices will be first verified.)
* Asthma, injuries, or other health conditions which inhibit daily physical activity
* Subjects must not already meet the recommended amount of physical activity of moderate-intensity physical activity for 150 minutes a week or 75 minutes at vigorous-intensity a week.
* Duke students are excluded from this study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity as measures by FitBit | Baseline (14 days after the 1st visit), End of study (80 days after the MR visit)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Samanez-Larkin, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No